CLINICAL TRIAL: NCT05764538
Title: DAOIB for the Treatment of Cognitive Impairment Induced by COVID-19 -An Open Trial
Brief Title: DAOIB for the Treatment of Brain Fog
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200988A3
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAOIB (Experimental)
  Interventions: Drug: DAOIB

INTERVENTIONS:
Drug: DAOIB — The DAOIB dose will be adjusted every 8 weeks according to clinical evaluation

SUMMARY:
This is a 24-week open trial. We will enroll long-COVID patients with cognitive impairments. All patients will receive DAOIB for 24 weeks. We will assess the patients every 8 weeks during the treatment period (weeks 0, 8, 16, and 24). We hypothesize that DAOIB treatment will be beneficial in improving the cognitive function, mood symptoms, global functioning and quality of life in long-COVID patients with cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* "post-COVID-19 condition" defined by WHO (symptoms present at three months after SARS-CoV-2 infection and last for at least 2 months which cannot be explained by an alternative diagnosis)(Cabrera Martimbianco, Pacheco et al. 2021) and COVID-induced cognitive impairments
* physically healthy and have all laboratory assessments (including urine/blood routine, biochemical tests, and electrocardiograph) within normal limits
* have sufficient education to communicate effectively and are capable of completing the assessments of the study

Exclusion Criteria:

* history of significant cerebrovascular disease
* Hachinski Ischemic Score > 4
* major neurological, psychiatric or medical conditions other than long COVID-induced cognitive impairments
* memantine use (memantine is an NMDAR partial antagonist)
* substance (including alcohol) abuse or dependence
* delusion, hallucination or delirium symptoms
* severe visual or hearing loss
* inability to follow the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale scores range from 0 (best) to 70 (worst)

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The assessment appears to be a suitable instrument for evaluating activities of daily living in early-phase dementia. Its scores range from 0 (worst) to 78 (best)
Change from baseline in Quality of life score at week 8, 16 and 24 | week 0, 8, 16, 24
  Quality of life will be assessed by Medical Outcomes Study Short-Form-36 (SF-36). The SF-36 consists of eight sections: (1) vitality, (2) physical functioning, (3) bodily pain, (4) general health perceptions, (5) physical role functioning, (6) emotional role functioning, (7) social role functioning, and (8) mental health.
Change from baseline of 17-item Hamilton Rating Scale for Depression | week 0, 8, 16, 24
  Assessment of depressive symptoms. The 17-item Hamilton Rating Scale for Depression will be measured every 8 weeks
Change from baseline of Hamilton Anxiety Rating Scale | week 0, 8, 16, 24
  Assessment of anxiety symptoms. The Hamilton Anxiety Rating Scale will be measured every 8 weeks
Change from baseline of Perceived Stress Scale | week 0, 8, 16, 24
  Assessment of stress and anxiety symptoms. The Perceived Stress Scale will be measured every 8 weeks
Change from baseline in the score of a battery of additional cognitive tests | week 0, 8, 16, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (Wechsler Memory Scale, Spatial Span), verbal/nonverbal learning and memory tests (Wechsler Memory Scale, Word Listing)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No